CLINICAL TRIAL: NCT00403975
Title: A Multi-Center, Parallel Group, Double-Masked, Randomized, Placebo-Controlled Study of Multiple Ocular Instillations of Diquafosol Tetrasodium Ophthalmic Solution, 2% in Subjects With Dry Eye Disease
Brief Title: Study of Diquafosol Tetrasodium Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-109
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: diquafosol tetrasodium ophthalmic solution, 2%

SUMMARY:
The purpose of this trial is to assess the effectiveness and safety of 2% diquafosol tetrasodium ophthalmic solution versus placebo following 6 weeks of treatment in subjects with mild to moderate dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity in both eyes of at least +0.7
* six-month documented history of dry eye disease
* as least mild severity in 1 of the 5 dry eye symptoms
* corneal fluorescein staining of greater than or equal to 3 and less than or equal to 6 (out of 15)

Exclusion Criteria:

* permanent conjunctival goblet cell loss or scarring conditions
* ongoing contact lens wear
* current topical ophthalmic medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change in dry eye testing measures

SECONDARY OUTCOMES:
Change in dry eye testing measures and symptoms